CLINICAL TRIAL: NCT02108184
Title: Comparison of the Eradications Rates of Sequential Therapy Versus Concomitant Therapy of Treatment of Helicobacter Pylori Infection in Korea
Brief Title: Comparison of the Eradications Rates of Sequential Therapy Versus Concomitant Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sung min, Park, fellow, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSungmin
Record Dates: First submitted 2014-02-26; First posted 2014-04-09 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter eradication rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sequential therapy 10 days (Experimental): 1.(pantoprazole 40 mg + amoxicillin 1.0 g bid) for the first 5 days, subsequently (pantoprazole 40 mg + clarithromycin 500 mg + metronidazole 500 mg bid) for the next 5 days
  Interventions: Drug: Sequential therapy 10 days
- Sequential therapy 14 days (Active Comparator): (pantoprazole 40 mg + amoxicillin 1.0 g bid) for the first 7days, subsequently (pantoprazole 40 mg + clarithromycin 500 mg + metronidazole 500 mg bid) for the next 7 days
  Interventions: Drug: Sequential therapy 14 days
- Concomitant therapy 10 days (Active Comparator): (pantoprazole 40 mg + amoxicillin 1.0 g + clarithromycin 500 mg + metronidazole 500 mg bid) for 10 days
  Interventions: Drug: Concomitant therapy 10 days
- Concomitant therapy 14 days (Active Comparator): (pantoprazole 40 mg +amoxicillin 1.0 g + clarithromycin 500 mg + metronidazole 500 mg bid) for 14 days
  Interventions: Drug: Concomitant therapy 14 days

INTERVENTIONS:
Drug: Sequential therapy 10 days — (pantoprazole 40 mg + amoxicillin 1.0 g) bid for the first 5 days, subsequently (pantoprazole 40 mg + clarithromycin 500 mg + metronidazole 500 mg ) bid for the next 5 days : Sequential therapy 1
  Arms: Sequential therapy 10 days
Drug: Sequential therapy 14 days — (pantoprazole 40 mg + amoxicillin 1.0 g bid) for the first 7days, subsequently (pantoprazole 40 mg + clarithromycin 500 mg + metronidazole 500 mg bid) for the next 7 days : Sequential therpay 2
  Arms: Sequential therapy 14 days
Drug: Concomitant therapy 10 days — (pantoprazole 40 mg + amoxicillin 1.0 g + clarithromycin 500 mg + metronidazole 500 mg ) bid for 10 days : Concomitant therapy 1
  Arms: Concomitant therapy 10 days
Drug: Concomitant therapy 14 days — (pantoprazole 40 mg +amoxicillin 1.0 g + clarithromycin 500 mg + metronidazole 500 mg bid) for 14 days : Concomitant therapy 2
  Arms: Concomitant therapy 14 days

SUMMARY:
Comparison of the eradications rates of sequential therapy versus concomitant therapy of treatment of Helicobacter pylori infection in Korea.

single center, randomized trial

1. (pantoprazole 40 mg + amoxicillin 1.0g + clarithromycin 500 mg + metronidazole 500 mg) twice for 10 days
2. (pantoprazole 40 mg + amoxicillin 1.0g + clarithromycin 500 mg + metronidazole 500 mg) twice for 14 days
3. (pantoprazole 40 mg + amoxicillin 1.0g) twice for 5 days and subsequent pantoprazole 40mg + clarithromycin 500 mg + metronidazole 500 mg) twice for 5 days
4. (pantoprazole 40 mg + amoxicillin 1.0g) twice for 7 days and subsequent pantoprazole 40mg + clarithromycin 500 mg + metronidazole 500 mg) twice for 7 days

1st endpoint : Helicobacter pylori eradication rates (intention to treatment, per-protocol) 2nd endpoint : adverse event(nausea, vomiting, dizziness, bitter sense) drug compliance

ELIGIBILITY:
Inclusion Criteria:

* 20~80 patients
* agreement of informed consent
* H.pylori positive (biopsy, CLO)
* Peptic ulcer disease, mucosa associated lymphoid tissue lymphoma, Post endoscopic submucosal dissection status due to early gastric cancer

Exclusion Criteria:

* H.pylori eradication history
* severe hepatic, renal, cardiac failure
* pregnancy, participant of other study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of the eradications rates of sequential therapy versus concomitant therapy of treatment of Helicobacter pylori infection in Korea. | required average 10 weeks to assess Helicobacter pylori eradication rate from 1st visit
  To assess Helicobacter pylori eradication rates

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St.Mary hospital, Incheon, Bupyung, South Korea

REFERENCES:
- [Background] Lim JH, Lee DH, Choi C, Lee ST, Kim N, Jeong SH, Kim JW, Hwang JH, Park YS, Lee SH, Shin CM, Jo HJ, Jang ES, Song Is, Jung HC. Clinical outcomes of two-week sequential and concomitant therapies for Helicobacter pylori eradication: a randomized pilot study. Helicobacter. 2013 Jun;18(3):180-6. doi: 10.1111/hel.12034. Epub 2013 Jan 11. PMID 23305083
- [Result] Kim JS, Kim BW, Ham JH, Park HW, Kim YK, Lee MY, Ji JS, Lee BI, Choi H. Sequential Therapy for Helicobacter pylori Infection in Korea: Systematic Review and Meta-Analysis. Gut Liver. 2013 Sep;7(5):546-51. doi: 10.5009/gnl.2013.7.5.546. Epub 2013 Aug 14. PMID 24073312